CLINICAL TRIAL: NCT06023394
Title: Laryngeal Mask Airway Versus Endotracheal Intubation for Laparoscopic Inguinal Hernia Repair
Brief Title: Laryngeal Mask Airway in Laparoscopic Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Emily Weisberg, Physican, M.D., Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Study00002580
Record Dates: First submitted 2023-08-04; First posted 2023-09-05 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Inguinal Hernia; Inguinal Hernia, Indirect; Inguinal Hernia Bilateral; Inguinal Hernia Unilateral
MeSH Terms: conditions — Hernia, Inguinal | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort A: Receives Laryngeal Mask Airway Device (Other): In this study arm, after induction of general anesthesia, the patients will receive a laryngeal mask airway device.
  Interventions: Device: Laryngeal Mask Airway
- Cohort B: Receives Endotracheal Tube Device (Other): In this arm, after induction of general anesthesia, the patients will receive an endotracheal tube airway device.
  Interventions: Device: Endotracheal Tube Device

INTERVENTIONS:
Device: Laryngeal Mask Airway — Laryngeal mask airway will be used as an airway device for Cohort A in the standard fashion.
  Arms: Cohort A: Receives Laryngeal Mask Airway Device
Device: Endotracheal Tube Device — Endotracheal tube airway will be used as an airway device for Cohort B in the standard fashion.
  Arms: Cohort B: Receives Endotracheal Tube Device

SUMMARY:
This prospective randomized study will evaluate the effectiveness of laryngeal mask airway (LMA) versus endotracheal intubation (ETT) for patients undergoing laparoscopic inguinal hernia at CMH.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness during general anesthesia of laryngeal mask airway versus endotracheal tube for laparoscopic inguinal hernia repair. There are limited pediatric literature evaluating the use of laryngeal mask airway for laparoscopic procedures compared with traditional endotracheal intubation. This study aims to add to this literature in providing information comparing the two techniques. The rationale for this study is to show that general anesthesia with laryngeal mask airway is an effective and non-inferior technique compared with general anesthesia with endotracheal intubation in pediatric patients undergoing laparoscopic inguinal hernia repair and may offer benefits in terms of efficiency of care and respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic inguinal hernia repair.
* Ages 12 months to 8 years of age
* American Society of Anesthesiologists Physical Status Classification ASA 1 or 2
* ASA 1- A normal, healthy patient
* ASA 2- A patient with mild systemic disease
* Elective with appropriate NPO status
* English speakers
* Spanish speakers

Exclusion Criteria:

* Patients with current gastroesophageal reflux
* Obesity (CDC >= 95th %ile)
* Contraindications to study protocol medications

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weisberg EL, Pieters BJ, Elman MS, Nonnemacher CJ, Noel-MacDonnell J, Oyetunji TA. The Use of Laryngeal Mask Airway Versus Endotracheal Intubation in Pediatric Laparoscopic Inguinal Hernia Repair: A Randomized Controlled Trial. J Pediatr Surg. 2025 Aug;60(8):162367. doi: 10.1016/j.jpedsurg.2025.162367. Epub 2025 May 15. PMID 40381798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
Started | 31 | 31
Completed | 25 | 25
Not Completed | 6 | 6
Not completed — Surgery was not performed laparoscopically | 4 | 2
Not completed — Surgery not performed (hernia not identified on diagnostic laparoscopy) | 0 | 3
Not completed — Did not receive allocated intervention (Patient received ETT per surgeon) | 1 | 0
Not completed — Did not received allocated intervention (no airway device documented in EMR) | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.5 [2 to 5.4] | 3.1 [2.2 to 4.8] | 3.21 [2.01 to 4.95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 18 | 19 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation Measured by Pulse Oximetry in Percent Saturation
Description: Oyxgen saturation will be measured by pulse oximetry in percent saturation at three time points during the anesthetic
Time Frame: Patients will have oxygen saturation measured directly after placement airway device, the first oxygen saturation recorded five minutes after the start of surgery, and immediately prior to removal airway device, assessed up to 2 hours.
Measure: Median (Inter-Quartile Range); unit: Percent Saturation
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
Number analyzed (Participants) | 25 | 25
Percent Saturation
  SpO2 after placement airway device | 100 [100 to 100] | 100 [99 to 100]
  SpO2 5 minutes after surgery start | 100 [100 to 100] | 100 [99 to 100]
  SpO2 prior to airway device removal | 100 [100 to 100] | 100 [99 to 100]

2. Secondary Outcome: End-tidal Carbon Dioxide Measured by Capnography in mm Hg
Description: Patients will have end-tidal carbon dioxide measured by capnography in mm Hg at three standardized time points during anesthesia.
Time Frame: Patients will have end-tidal carbon dioxide measured directly after placement of device, the first end-tidal carbon dioxide measurement recorded five minutes after the start of surgery, and immediately prior to removal of device, assessed up to 2 hours.
Measure: Median (Inter-Quartile Range); unit: millimeters mercury (mm Hg)
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
Number analyzed (Participants) | 25 | 25
millimeters mercury (mm Hg)
  ETCO2 after placement of airway device | 44 [39 to 50] | 43 [41 to 48]
  ETCO2 5 minutes after surgery start | 47 [43 to 49] | 48 [42 to 50]
  ETCO2 prior to removal of airway device | 45 [43 to 53] | 49 [43 to 57]

3. Secondary Outcome: Peak Airway Pressure Will be Measured in cm H2O
Description: Patients will have peak airway pressure in cm H2O measured at three standardized time points during anesthesia.
Time Frame: Patients will have peak airway pressure measured directly after placement airway device, the first airway pressure recorded five minutes after the start of surgery, and immediately prior to removal airway device, assessed up to 2 hours.
Measure: Median (Inter-Quartile Range); unit: cm H20
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
Number analyzed (Participants) | 25 | 25
cm H20
  Peak airway pressure after placement of airway device | 11 [7 to 12] | 14 [12 to 16]
  Peak airway pressure 5 minutes after surgery start | 13 [11 to 14] | 16 [15 to 19]
  Peak airway pressure prior to removal of airway device | 7 [1 to 11] | 11 [5 to 14]

4. Secondary Outcome: Documentation of Laryngospasm Occurrence
Description: Will document if laryngospasm occurs in both groups at any time during the surgery.
Time Frame: Patients will have the occurrence of laryngospasm documented at any time point during the surgery, assessed up to 2 hours.
Measure: Number; unit: Presence of laryngospasm
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
Number analyzed (Participants) | 25 | 25
Presence of laryngospasm | 0 | 0

5. Secondary Outcome: Documentation of Oxygen Desaturation
Description: Will document if oxygen desaturation occurs at any time during the surgery as defined as an oxygen saturation of less than 90%.
Time Frame: Patients will have the occurrence of oxygen desaturation documented if it occurs at any time point during the surgery, assessed up to 2 hours.
Measure: Number; unit: Occurence of oxygen desaturation
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
Number analyzed (Participants) | 25 | 25
Occurence of oxygen desaturation | 1 | 1

ADVERSE EVENTS:
Time Frame: During anesthetic time, defined as induction of anesthesia, to time of LMA or ETT removal documented by the anesthesia time, assessed up to 2 hours.
Arm/Group | Cohort A: Receives Laryngeal Mask Airway Device | Cohort B: Receives Endotracheal Tube Device
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT06023394/Prot_SAP_000.pdf